CLINICAL TRIAL: NCT04783259
Title: Exploring the Views of Medical Students on Medical Escape Room Experiences With Narrow Learning Objectives and Structured Debriefings
Brief Title: Structured Debriefings After Medical Escape Rooms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Tami Jørgensen, Medical student, Copenhagen Academy for Medical Education and Simulation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Debriefing MERGE
Record Dates: First submitted 2021-02-22; First posted 2021-03-05 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Interactive Teaching
Keywords: Escape room; Debriefing; Structured; Learning goal; Learning objective

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Structured approach — Structured approach with a narrow learning objective. The structured approach concerns a pre-escape room lecture and post-escape room debriefing
  Other Names: Narrow learning objective

SUMMARY:
An escape room is a game-like experience, where participants solve a series of logic based puzzles. Such game-like experiences are being increasingly used in the educations of medical professionals. With this research project, the researchers aim to explore medical students' experiences and perceived learning outcome of narrow learning objectives in a medical escape room experience. The learning experience will be structured with a short lecture, focussed instructions, a medical escape room scenario and a structured debriefing. The aim is that the study will create the foundation for general principles for the conduct of medical escape room experiences.

DETAILED DESCRIPTION:
Introduction

Background

Current medical students prefer innovative and interactive education styles such as gamification. Gamification concerns the act of applying game mechanics to a non-gaming environment, e.g. by putting themes of a clinical situation in the frames of a game. This concept is being increasingly frequently used in the education of healthcare professionals, and studies have shown that it appears to be effective to reach the learning outcome. In the study "Priming healthcare students on the importance of non-technical skills in healthcare: How to set up a medical escape room game experience" by Rosenkrantz et al. 2019, a medical escape room was designed to raise awareness about non-technical skills (NTS) among healthcare professionals. The escape room was named Medical Escape Room Gaming Experience (MERGE). As with other common escape rooms, MERGE was designed as a game like exercise with puzzles, which in this room were medical-themed. However, the primary focus is not the medical technical skills, and thus the puzzles are mainly logic-based with a medical twist. This is to keep focus on developing NTS.

Game-like exercises, like MERGE, tend to have a complexity that allows addressing many different learning goals, depending onto what the attention is guided by the educator. In the researchers' experience, often a broad learning goal is initiated by a rather general instruction to pay attention e.g. to the "non-technical skills" or to "communication". This enables many possible discussions, also taking the interest of participants into account. The downside can be that the discussion might be superficial and erratic, as conflicting interests in the group might lead to frequent changes in topics. Another approach is to specify some narrow learning objectives in more detail, e.g. "identify the different sources of information", directing the discussion on very specific aspects of the scenario. This entails that potentially a lot of interesting elements remain uncovered, and that participants might not get the chance to discuss what they think is most important for them. On the other hand, the discussion of the learning objectives can reach deeper reflection levels, as fewer topics need to be covered and as less time is used to coordinate what should be discussed.

Rosenkrantz et al. and several others have proposed that the participants of an escape rooms experiences may achieve a greater learning outcome if they are debriefed by a trained professional after participating in the escape room. The trained debriefer can also be a peer to the learners. Peer-to-peer feedback is suggested to have a positive effect on learning outcome. Debriefing can be defined as the act of reviewing critical actions that unfolded during the course of a simulation scenario, and in its form, it is conversational, bidirectional, interactive, and reflective. Debriefing is known to enhance the learning outcome by allowing for reflection on educational experiences. Several experiments with debriefing after medical escape rooms have been carried out in the last few years. However, only the studies by Friedrich et al. and the two studies by Zhang et al. had the aspect of debriefing as a point of focus. In these three studies, the participants answered different questionnaires, where some of the questions regarded the debriefing. All three studies concluded that the participants appreciated the post-escape room debriefing. In addition, the studies by Zhang et al. concluded that the participants would have preferred a more structured debriefing session to help them analyse aspects of communication and problem-solving. All of the aforementioned studies with post-escape room debriefing had broad learning objectives primarily concerning communication. No studies concerning medical escape rooms have evaluated the use of narrow learning objectives in a medical escape room.

Aims

With this research project, the researchers aim to explore the participants' experiences and perceived learning outcome of narrow learning objectives in a medical escape room experience. The learning experience will be structured with a short lecture, focussed instructions, the MERGE scenario and a structured debriefing. The aim is that the study will create the foundation for general principles for the conduct of medical escape room experiences.

Method

This is an explorative qualitative intervention study. A qualitative, summarising approach is used to analyse responses to the intervention. We will achieve this by exploring participants' experiences shortly after they have undergone a structured post-escape room debriefing. The aforementioned escape room, MERGE, will be conducted with teams of medical students.

Design

Before the escape room begins, the participants will participate in a brief video recorded lecture by a medical student concerning the learning objectives. Afterwards, the facilitator will brief the participants about the voluntary nature of their participation in the study, and the learning objectives of the escape room. These measures are thought to establish a common ground for the discussion in the debriefing. When the participants have finished the escape room by completing all the riddles, they will be taken to an adjacent room. Here, an educator, a person other than the facilitator, will debrief them. The debriefing will follow a manual, but the educator will have observed the participants through the see-through mirror in order to guide the group in their individual debriefing. Afterwards, the educator will leave, and an interviewer will join the group and ask them a series of standardised questions regarding the escape room gaming experience and the following debriefing. Lastly, the participants will answer a questionnaire regarding, age, gender, and their experience related to simulation, debriefing, etc. As all the participants will be Danish speaking, the language for both the escape room, the debriefing, the interview and the questionnaire will be in Danish.

Participants and sample size

The participants of this study will be medical students who have completed the fourth year of their studies at the University of Copenhagen in Denmark (UCPH). At this point in their studies, they have completed four months of internship, experiencing the clinical practice of young doctors. As a group, they have little experience with simulation, but everyone will have tried it a few times. The recruitment of the participants will be executed by posting a notice on a social media platform, including the vast majority of medical students at UCPH. The participants are to apply as premade groups of four to five people, and the applicants will be chosen based on the order in which they apply.

The goal is to conduct eight to ten sessions of the escape room with groups of four to five participants each, and participants will only be allowed to participate once. The study group estimates that this is the number of simulations required to receive sufficient qualitative data. The researchers will check for data saturation during the analysis, which they expect will be reached after about six sessions. In case saturation is not reached after all ten sessions, further sessions will be conducted until saturation is reached.

The Intervention

The intervention in this study is a structured experiential learning session including a short video lecture, focussed instructions, the MERGE scenario, and a structured standardized four-layered post session debriefing with narrow learning objectives. The video lecture will concern the learning objectives and will be developed within the research team and recorded with a medical student delivering it. Also the focussed instructions will be developed within the research team and delivered by the facilitator, who also conducts the MERGE session. The debriefing of the participants will be a semi-structured conversation lead by an educator. The educator will be a medical student practical experience in peer-to-peer debriefing of medical students after medical simulations. The debriefing will have a narrow focus, revolved around two learning objectives. Rosenkrantz et al. 2019 suggested that the NTS concerning information gathering and exchange are the most viable of being focus points in the MERGE. Therefore, the learning objectives of focus in the debriefing will be: "Recognising the different ways of exchanging information" and "Discussing the impact of exchanging information on problem-solving". These learning objectives are designed to explore the exchange of information on several of Bloom's taxonomical levels. The first learning objective concerns knowledge and comprehension, and the second concerns application and analysis. The educator will guide the conversation using the manual shown below. The manual follows the common four-phase debriefing model inspired by Steinwach 1992 and PEARLS. First, the educator sets the scene by explaining the course of the debriefing. The debriefing then starts with a reaction phase, where the participants are encouraged to express their feelings and ask any technical questions they may have regarding the escape room. This is followed by a focused description phase, where the participants discuss the first learning objective by describing the different ways they exchanged information during the escape room. Hereafter comes the analysis phase, during which the second learning objective concerning the impact of exchanging information is explored and discussed. Lastly, the debriefing is rounded off in the application phase, where the participants transfer the events of the simulation to clinical practice and sum up the key learning points. As the debriefing is a semi-structured conversation, the manual is not expected to be followed meticulously regarding the order of the points. However, all the points must be covered, and the overall structure with the four phases should be maintained in all concerns.

The manuscript for the educator

0. Setting the scene (2 min)

• "In this debriefing, we are going to reflect on your experiences. It will take about 45 minutes. We will first discuss shortly, what happened in the escape room. Then we are all going to reflect on how you shared information. Lastly, we will look at what you can take with you."

1. Reaction

   * "How are each of you feeling right now?"
   * "Are you sitting with any technical questions about the riddles or the escape room in general at this moment?"
   * "Now then, having answered your questions, I am going to continue with the debriefing."
2. Description

   * "We are - in this debriefing - especially interested in how you shared information with each other. We could discuss many things, but we would like to focus on this aspect."
   * "I want each of you to answer the question: 'What were the different ways you used to exchange information?' I want you to describe how you did it in as much detail as possible." Start with one and then ask the others for additions. Consider taking notes that all can see.
   * If you noticed any additional examples of information exchange, lead their attention to it and make them describe it by saying something like: "I also noticed a point where … can you elaborate what happened there?"
3. Analysis

   * "What went well in today's game in regards to the exchange of information, and how did it affect your performance in the escape room?"
   * "How and why would the progression have been different if you had not been allowed to talk to each other?"
   * "Were there phases of the escape room, where the exchange of information was more or less important? Please elaborate."
   * "Did you experience any situations where you found it difficult to exchange information with a member of your team? When and why?"
   * "How could you have optimised your exchange of information?"
4. Application

   * "How can the things you learned today be applied in your clinical practice?"
   * "Lastly, I want each of you to mention the most important thing that you learned from today's events."

Assessment of the intervention: Semi-structured interviews

The interview of the participants will be a semi-structured group interview concerning the participants' perceived value of medical escape rooms and the following debriefing, and their opinions about the narrow learning objectives. The interview will follow the questions shown below. The interview will be video and audio recorded as material for the following analysis.

Questions

The escape room

• "How was your experience with the escape room? Is there anything you want to emphasise?"

The debriefing

* "What do you think about the debriefing?"
* "What are the pros and cons of a structured debriefing like you had versus a different format, e.g. an unstructured conversation?"
* "Would you have preferred that the format had been less structured? Why/ why not?"
* "How do you feel about the very narrow focus of the debriefing, i.e. the exchange of information?"
* "Were there any topics that you wanted to discuss, but couldn't due to the narrow learning objective?"
* "Would you rather have had more time to discuss certain aspects?
* After your considerations in this interview, I ask again: what do you think about the debriefing?

The learning outcome

* "When during the escape room and/or debriefing do you feel that you learned something concerning exchange of information?"
* "Did you learn anything besides exchange of information? What and when?"
* "Do you experience that the debriefing has affected your learning outcome today? How and why?"

Analysis of debriefings and interviews

The interviews will provide data for analysis in the form of video and audio recordings. These data will be analysed using systematic text condensation. First, the recordings of the interviews from the first six escape rooms will be transcribed. These transcripts will then be coded in a condensating fashion and any relevant key points will be identified. Afterwards, the researchers will watch the recordings of the remaining interviews, focusing on whether they provide any new inputs or whether saturation has been achieved. Any of these will then be transcribed and coded as well, should they provide new inputs. The codes will be grouped in order to create themes, which will then be labelled by their common denominator. The themes and their connections will be described and discussed. Based on this discussion, the researchers will conclude how participants experience the learning setting and what kind of learning outcome they perceive. Based on the analysis of the participants' experiences, general principles for the conduct of medical escape room experiences will be derived.

ELIGIBILITY:
Inclusion Criteria:

* Medical students who have completed the fourth year of their studies at the University of Copenhagen in Denmark

Exclusion Criteria:

* Participants not available for the entire duration
* Symptoms indicating viral respiratory disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Condensed text categories | Within 1 year
  Debriefings and interviews will be transcribed and analysed by systematic text condensing. Major themes will be presented by occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Tami Jørgensen, bsc.med., Principal Investigator — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Academy of Medical Education and Simulation, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams NE. Bloom's taxonomy of cognitive learning objectives. J Med Libr Assoc. 2015 Jul;103(3):152-3. doi: 10.3163/1536-5050.103.3.010. PMID 26213509
- [Background] aSarage D, O'Neill BJ, Eaton CM. There is no I in Escape: Using an Escape Room Simulation to Enhance Teamwork and Medication Safety Behaviors in Nursing Students. Simulation & Gaming. 2020:1046878120976706.
- [Background] Eppich W, Cheng A. Promoting Excellence and Reflective Learning in Simulation (PEARLS): development and rationale for a blended approach to health care simulation debriefing. Simul Healthc. 2015 Apr;10(2):106-15. doi: 10.1097/SIH.0000000000000072. PMID 25710312
- [Background] Fanning RM, Gaba DM. The role of debriefing in simulation-based learning. Simul Healthc. 2007 Summer;2(2):115-25. doi: 10.1097/SIH.0b013e3180315539. No abstract available. PMID 19088616
- [Background] Felix HM, Beecham GB, Simon LV. Debriefing Theories and Philosophies in Medical Simulation. 2024 Sep 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551632/ PMID 31869096
- [Background] Friedrich C, Teaford H, Taubenheim A, Boland P, Sick B. Escaping the professional silo: an escape room implemented in an interprofessional education curriculum. J Interprof Care. 2019 Sep-Oct;33(5):573-575. doi: 10.1080/13561820.2018.1538941. Epub 2018 Oct 26. PMID 30362849
- [Background] Gentry SV, Gauthier A, L'Estrade Ehrstrom B, Wortley D, Lilienthal A, Tudor Car L, Dauwels-Okutsu S, Nikolaou CK, Zary N, Campbell J, Car J. Serious Gaming and Gamification Education in Health Professions: Systematic Review. J Med Internet Res. 2019 Mar 28;21(3):e12994. doi: 10.2196/12994. PMID 30920375
- [Background] Kinio AE, Dufresne L, Brandys T, Jetty P. Break out of the Classroom: The Use of Escape Rooms as an Alternative Teaching Strategy in Surgical Education. J Surg Educ. 2019 Jan-Feb;76(1):134-139. doi: 10.1016/j.jsurg.2018.06.030. Epub 2018 Aug 17. PMID 30126728
- [Background] Lerchenfeldt S, Mi M, Eng M. The utilization of peer feedback during collaborative learning in undergraduate medical education: a systematic review. BMC Med Educ. 2019 Aug 23;19(1):321. doi: 10.1186/s12909-019-1755-z. PMID 31443705
- [Background] McClarty KL, Orr A, Frey PM, Dolan RP, Vassileva V, McVay A. A literature review of gaming in education. Gaming in education. 2012:1-35.
- [Background] Moore K, Frazier RS. Engineering education for generation Z. American Journal of Engineering Education (AJEE). 2017;8(2):111-26.
- [Background] Nicholson S. Peeking behind the locked door: A survey of escape room facilities. Pozyskano z http://scottnicholson com/pubs/erfacwhite pdf. 2015.
- [Background] Rosenkrantz O, Jensen TW, Sarmasoglu S, Madsen S, Eberhard K, Ersboll AK, Dieckmann P. Priming healthcare students on the importance of non-technical skills in healthcare: How to set up a medical escape room game experience. Med Teach. 2019 Nov;41(11):1285-1292. doi: 10.1080/0142159X.2019.1636953. Epub 2019 Jul 23. PMID 31335239
- [Background] Sardi L, Idri A, Fernandez-Aleman JL. A systematic review of gamification in e-Health. J Biomed Inform. 2017 Jul;71:31-48. doi: 10.1016/j.jbi.2017.05.011. Epub 2017 May 20. PMID 28536062
- [Background] Schenarts PJ. Now Arriving: Surgical Trainees From Generation Z. J Surg Educ. 2020 Mar-Apr;77(2):246-253. doi: 10.1016/j.jsurg.2019.09.004. Epub 2019 Sep 24. PMID 31562032
- [Background] Shatto B, Erwin K. Teaching Millennials and Generation Z: Bridging the Generational Divide. Creat Nurs. 2017 Feb 1;23(1):24-28. doi: 10.1891/1078-4535.23.1.24. PMID 28196564
- [Background] Stewart LP. Ethical issues in postexperimental and postexperiential debriefing. Simul Gaming. 1992 Jun;23(2):196-211. doi: 10.1177/1046878192232007. No abstract available. PMID 11659673
- [Background] van Gaalen AEJ, Brouwer J, Schonrock-Adema J, Bouwkamp-Timmer T, Jaarsma ADC, Georgiadis JR. Gamification of health professions education: a systematic review. Adv Health Sci Educ Theory Pract. 2021 May;26(2):683-711. doi: 10.1007/s10459-020-10000-3. Epub 2020 Oct 31. PMID 33128662
- [Background] Zhang XC, Diemer G, Lee H, Jaffe R, Papanagnou D. Finding the 'QR' to Patient Safety: Applying Gamification to Incorporate Patient Safety Priorities Through a Simulated 'Escape Room' Experience. Cureus. 2019 Feb 5;11(2):e4014. doi: 10.7759/cureus.4014. PMID 31007972
- [Background] Zhang XC, Lee H, Rodriguez C, Rudner J, Chan TM, Papanagnou D. Trapped as a Group, Escape as a Team: Applying Gamification to Incorporate Team-building Skills Through an 'Escape Room' Experience. Cureus. 2018 Mar 2;10(3):e2256. doi: 10.7759/cureus.2256. PMID 29725559
- [Derived] Jorgensen T, Rosenkrantz O, Eberhard KE, Jensen TW, Dieckmann P. Perceptions of medical students on narrow learning objectives and structured debriefing in medical escape rooms: a qualitative study. BMC Med Educ. 2024 Apr 11;24(1):403. doi: 10.1186/s12909-024-05295-4. PMID 38605342